CLINICAL TRIAL: NCT06506331
Title: Impact of Preoperative Visceral Fat Area on Intraoperative Adverse Events in Patients Undergoing Laparoscopic Radical Gastrectomy: A Pooled Analysis From Two Randomized Trials
Brief Title: Impact of Preoperative VFA on Intraoperative Adverse Events in Patients Undergoing Laparoscopic Radical Gastrectomy
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Other Study IDs: 2024KY088
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; intraoperative adverse events; complications; visceral fat area; laparoscopic surgery
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high-VFA: VFA≥74 cm2
- low-VFA: VFA<74 cm2

SUMMARY:
Preoperative visceral fat area (VFA) is associated with an increased incidence of postoperative complications in gastric cancer (GC). However, the relationship between VFA and intraoperative adverse events (iAEs) remains unclear. Therefore, this study aimed to evaluate the impact of preoperative VFA on iAEs in patients undergoing laparoscopic radical gastrectomy for GC, using data from two prospective trials. Simultaneously, a predictive model for iAEs was constructed to provide a basis for the early identification of high-risk populations and the implementation of personalized perioperative management measures.

DETAILED DESCRIPTION:
A post hoc analysis was performed using data from two previous prospective studies ([NCT02327481] and [NCT01609309]). The patients were divided into high- and low-VFA groups. All iAEs were reviewed from the surgical videos and graded using ClassIntra. Logistic regression analyses were used for the construction of nomograms as predictive models.

ELIGIBILITY:
Inclusion Criteria:

This study comprised two prospective trials conducted at Fujian Medical University Union Hospital (FMUUH): the FUGES-001 study (ClinicalTrials.gov, NCT02327481) and a subset of the CLASS-01 multicenter study (ClinicalTrials.gov, NCT01609309)

Exclusion Criteria:

1. open surgery;
2. non-adenocarcinoma gastric cancers
3. Palliative surgery
4. Exploratory operation
5. CT data missing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A post hoc analysis was performed using data from two previous prospective studies ([NCT02327481] and [NCT01609309]).
Sampling Method: Non-Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
intraoperative adverse events(iAEs) | During surgery
  Intraoperative adverse events (iAEs) are important indicators for evaluating surgical quality and encompass a range of circumstances such as intraoperative bleeding, injury, and anesthesia-related events that may impact postoperative outcomes

SECONDARY OUTCOMES:
Postoperative complications | 30 days after surgery
  Postoperative complications were evaluated according to the Clavien-Dindo classification and categorized as surgical or medical

CONTACTS AND LOCATIONS:
Overall Officials: Changming Huang, PhD, Principal Investigator — Fujian Medical University Union Hospital

IPD SHARING:
Plan to Share IPD: No